CLINICAL TRIAL: NCT04402138
Title: Single Arm, Phase II Study of Acalabrutinib as Post-Autologous Blood or Marrow Transplant (BMT) Maintenance Therapy in Subjects With Mantle Cell Lymphoma
Brief Title: Treatment With Acalabrutinib Post Blood or Marrow Transplantation in Subjects With Mantle Cell Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: SCRI Development Innovations, LLC (Other)
Collaborators: Acerta Pharma, LLC (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LYM 155
Record Dates: First submitted 2020-05-15; First posted 2020-05-26 (Actual); Results first posted 2025-05-13 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Mantle Cell Lymphoma
Keywords: Acalabrutinib; Non Hodgkin's lymphoma; Blood or Marrow transplant; BMT; Maintenance therapy; Bruton's Tyrosine Kinase Inhibitor
MeSH Terms: conditions — Lymphoma, Mantle-Cell; Lymphoma, Non-Hodgkin | interventions — acalabrutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Acalabrutinib (Experimental): Acalabrutinib will be self-administered orally for up to approximately 2 years post-BMT.
  Interventions: Drug: Acalabrutinib

INTERVENTIONS:
Drug: Acalabrutinib — Acalabrutinib 129 mg will be self-administered orally twice daily (BID) starting from 100 day (+/- 7 days) Post-BMT on a 28-day schedule, with or without food, until the patient has reached approximately 2 years post-BMT.
  Other Names: Calquence

SUMMARY:
This is a phase II study to evaluate efficacy of Acalabrutinib as a maintenance therapy following blood or marrow transplant (BMT) in patients who have been diagnosed with mantle cell lymphoma.

DETAILED DESCRIPTION:
Mantle cell lymphoma (MCL) is one of approximately 100 different types of non-Hodgkin's lymphoma (NHL). Due to the aggressive and heterogeneous nature of MCL, majority of patients are diagnosed with advanced stage disease that requires immediate, diverse and aggressive courses of therapy to improve the outcome of the disease. The addition of blood or bone marrow transplantation (BMT) to the chemotherapy regimens is a critical factor to prolong duration of response in patients, however, the benefit of combination chemotherapy followed by BMT is often temporary as patients experience disease progression and mortality and this underscores the need for novel therapies as well as additional maintenance therapy strategies to prevent relapse post-BMT.

Acalabrutinib, a selective, irreversible small molecule inhibitor of Bruton's tyrosine kinase (BTK) is approved for the treatment of adult patients with MCL who have received at least 1 prior therapy

This study is a single arm, multi-center, phase 2 study of participants who will receive acalabrutinib as maintenance therapy post-BMT. Participants will undergo a standard of care BMT with conditioning regimen determined by the treating physician per institutional guidelines.The BMT procedure is not considered part of this study. Following completion of the BMT, maintenance therapy with acalabrutinib will begin on Day 100 in 28-day cycles. Participants will self-administer 129 mg acalabrutinib twice daily (BID) until they reach 2 years post-BMT (approximately 22 cycles). Participants will be followed for up to 5 years post-BMT for Progression Free Survival.

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria for Initial Enrollment (Screening #1):

Patients must meet all of the following criteria in order to be included in this research study:

1. Written informed consent, according to local guidelines, signed by the subject or by a legal guardian prior to the performance of any study-related screening procedures.
2. Men and women ≥18 years-of-age at the time of signature of the informed consent form (ICF).
3. A diagnosis of MCL confirmed by one of the following:

   * t(11;14) detected by fluorescence in situ hybridization (FISH), conventional cytogenetics, or other molecular evaluation
   * expression of cyclin D1 confirmed by immunohistochemistry.
4. Subject must have completed induction chemotherapy and plan to and be eligible to receive their first BMT per standard of care.
5. Availability of an archival paraffin-embedded tumor block for MRD testing.
6. The Investigator anticipates that the subject will meet the appropriate lab requirements listed in Screening #2 by Day 100.
7. Patients who received prior therapy with a BTK inhibitor are eligible to enroll.

Inclusion Criteria Post-BMT, Prior to Day 100 (Screening #2):

1. Adequate organ system function defined as:

   * Absolute neutrophil count (ANC) ≥1,000/mm3.
   * Total bilirubin ≤1.5 x the upper limit of normal (ULN) (except for previously documented Gilbert's syndrome)
   * Platelet count ≥75,000/mm3. Platelet infusions to meet eligibility criteria are not allowed within 3 days of study enrollment.
   * Alanine aminotransferase (ALT)/aspartate aminotransferase (AST) ≤2.5 x ULN
   * Calculated creatinine clearance (CrCl) ≥30 mL/min as calculated by the CockcroftGault method. Estimated CrCl (glomerular filtration rate [GFR]) = (140-age [years]) x (weight [kg]) x Fa /(72 x serum creatinine [mg/dL]) a where F = 0.85 for females and F = 1 for males
2. Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, or 2.
3. Subjects who did not receive an anti-cancer therapy (including surgery, radiotherapy, chemotherapy, immunotherapy, or investigational therapy) during the time between their transplant and the start of study therapy. Subjects must have recovered (e.g., Grade ≤1 or baseline) from AEs associated with prior cancer therapy. Note: Subjects with Grade ≤2 neuropathy or Grade ≤2 alopecia are an exception to the latter criterion and may qualify for the study.
4. Woman of childbearing potential (WoCBP) who are sexually active with male partners must use highly effective methods of contraception during treatment and for 2 days after the last dose of acalabrutinib. For male subjects with a pregnant or non-pregnant WoCBP partner, no contraception measures are required. A WoCBP must have a negative pregnancy test (urine or serum) at the time of screening and 72 hours before starting the study drug or have evidence of non-childbearing potential by fulfilling one of the following criteria:

   * Post-menopausal women, defined as either women aged >50 years and amenorrheic for ≥12 months following cessation of all exogenous hormonal treatments or women <50 years old who have been amenorrheic for ≥12 months following the cessation of exogenous hormonal treatments, and have serum follicle- stimulating hormone (FSH) and luteinizing hormone (LH) levels in the post- menopausal range for the institution.
   * Documentation of irreversible surgical sterilization by hysterectomy, bilateral oophorectomy or bilateral salpingectomy, but not tubal ligation
   * Medically confirmed, irreversible premature ovarian failure.
5. Willing and able to participate in all required evaluations and procedures in this study protocol including swallowing capsules without difficulty.
6. Ability to understand the purpose and risks of the study and provide signed and dated informed consent and authorization to use protected health information (PHI).

Exclusion Criteria:

Patients who meet any of the following criteria will be excluded from study entry:

1. Subjects who have relapsed or progressed at any time prior to BM
2. Subjects with known mutations that confer resistance to a BTK inhibitor.
3. Confirmed clinical PD since the time of BMT
4. Prior malignancy (or any other malignancy requiring active treatment), except for adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, or other cancer from which the subject has been disease free for ≥2 years or that will not limit survival to <2 years. The exceptions are:

   * Subjects treated with curative intent >2 years prior to enrollment and have a low probability of recurrence.
5. Clinically significant cardiovascular disease such as uncontrolled or symptomatic arrhythmias, congestive heart failure, or myocardial infarction within 6 months of screening, or any Class 3 or 4 cardiac disease as defined by the New York Heart Association Functional Classification.
6. Malabsorption syndrome, disease significantly affecting gastrointestinal function, resection of the stomach or small bowel that is likely to affect absorption, symptomatic inflammatory bowel disease, partial or complete bowel obstruction, or gastric restrictions and bariatric surgery, such as gastric bypass.
7. Known history of infection with human immunodeficiency virus (HIV) or any uncontrolled active systemic bacterial, fungal, parasitic or viral infection. Infections are considered controlled if appropriate therapy has been instituted and, at the time of screening, no signs of infection progression are present.
8. Known history of drug-specific hypersensitivity or anaphylaxis to study drug (including active product or excipient components).
9. Active bleeding or history of bleeding diathesis (e.g., hemophilia or von Willebrand disease).
10. Uncontrolled autoimmune hemolytic anemia or idiopathic thrombocytopenic purpura.
11. Requires treatment with a strong CYP3A4 inhibitor/inducer
12. Requires or is receiving anticoagulation treatment with warfarin or equivalent vitamin K antagonists (e.g., phenprocoumon) within 7 days of first dose of study drug.
13. Prothrombin time (PT)/ international normalized ratio (INR) or activated partial thromboplastin time (aPTT) >2 x ULN (in the absence of lupus anticoagulant).
14. Requires treatment with proton-pump inhibitors (e.g., omeprazole, esomeprazole, lansoprazole, dexlansoprazole, rabeprazole, or pantoprazole). Subjects receiving proton pump inhibitors who switch to H2-receptor antagonists or antacids are eligible for enrollment to this study.
15. History of significant cerebrovascular disease/event, including stroke or intracranial hemorrhage, within 6 months before the first dose of study drug.
16. Major surgical procedure within 28 days of first dose of study drug. Note: If a subject had major surgery, they must have recovered adequately from any toxicity and/or complications from the intervention before the first dose of study drug.
17. Hepatitis B or C serologic status: subjects who are hepatitis B core antibody (anti-HBc) positive and who are hepatitis B surface antigen (HbsAg) negative will need to have a negative PCR result. Those who are HbsAg positive or hepatitis B PCR positive will be excluded. Subjects who are hepatitis C antibody positive will need to have a negative PCR result. Those who are hepatitis C PCR positive will be excluded.
18. Breastfeeding or pregnant.
19. Concurrent participation in another therapeutic clinical trial.
20. Psychological, familial, sociological, or geographical conditions that do not permit compliance with the protocol and/or follow-up procedures outlined in the protocol.
21. The inability to swallow capsules.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2020-08-07 (Actual); Primary Completion 2024-04-05 (Actual); Study Completion 2024-04-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Tees, MD, Study Chair — Colorado Blood Cancer Institute
Locations (4):
- United States (4):
  - Colorado Blood Cancer Institute, Denver, Colorado
  - Tulane University, Office of Clinical Research, New Orleans, Louisiana
  - HCA Midwest, Kansas City, Missouri
  - Tennessee Oncology, Nashville, Tennessee

RESULTS

PARTICIPANT FLOW:
Groups:
- Acalabrutinib: Acalabrutinib will be self-administered orally for up to approximately 2 years post-BMT.
  Acalabrutinib: Acalabrutinib 129 mg BID will be self-administered orally starting from 100 day (+/- 7 days) Post-BMT on a 28-day schedule, with or without food, until the patient has reached approximately 2 years post-BMT.
Period: Overall Study
Arm/Group | Acalabrutinib
Started | 15
Completed | 12
Not Completed | 3
Not completed — Progressive Disease | 2
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Groups:
- Acalabrutinib: Acalabrutinib will be self-administered orally for up to approximately 2 years post-BMT.
  Acalabrutinib: Acalabrutinib 129 mg BID will be self-administered orally starting from 100 day (+/- 7 days) Post-BMT on a 28-day cycle schedule, with or without food, until the patient has reached 2 years post-BMT.
Arm/Group | Acalabrutinib
Number analyzed (Participants) | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 6
  >=65 years | 9
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 11
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 12
  More than one race | 0
  Unknown or Not Reported | 3
Region of Enrollment [Number; unit: participants]
  United States | 15

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival Rate (PFS) at 2 Years Post-Blood or Marrow Transplant (BMT)
Description: Progression Free Survival Rate is defined as the Kaplan-Meier estimate of the percentage of participants who are alive and free of disease progression according to Response Evaluation Criteria in Lymphoma (RECIL 2017) for up to 2 years post-BMT.
  According to RECIL, disease progression is defined as following criteria: >20% increase in sum of longest diameters of target lesions, for small lymph nodes measuring <15 mm post therapy, a minimum absolute increase of 5 mm and the longest diameter should exceed 15mm, or appearance of new lesions.
Time Frame: 2 years after date of BMT procedure for each patient
Population: Participants who receive at least one dose of acalabrutinib, who have an adequate baseline disease assessment and an adequate post-baseline assessment, or those who discontinue due to death or PD prior to their first assessment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Acalabrutinib
Number analyzed (Participants) | 15
percentage of participants | 73.5 [35.9 to 91.1]

2. Secondary Outcome: Conversion Rate From Minimal Residual Disease Positive (MRD+) to Minimal Residual Disease Negative (MRD-)
Description: Percentage of participants whose whole blood or bone marrow results transition from MRD positive before study treatment to MRD negative at 2 years post-BMT. An MRD negative status will be defined as all results from whole blood and bone marrow that are negative for the presence of residual clonal cells (with assay sensitivity of 10^-6) per Adaptive Biotechnologies' reporting methods.
Time Frame: Assessed at day 100 post-BMT procedure (prior to beginning maintenance treatment with study drug) and 2 years post-BMT
Population: Participants who received one dose of study drug and had post-BMT MRD tested
Measure: Number; unit: percentage of participants
Arm/Group | Acalabrutinib
Number analyzed (Participants) | 15
percentage of participants | 13.3

3. Secondary Outcome: Minimal Residual Disease (MRD) Correlation With Progression Free Survival (PFS)
Description: To compare the Kaplan-Meier estimated PFS rate for MRD negative population with MRD positive population. Progression-free survival is defined as the time from date of BMT procedure (day 0) until the date of objective radiological PD according to Response Evaluation Criteria in Lymphoma (RECIL 2017) or death. According to RECIL, disease progression is defined as following criteria: >20% increase in sum of longest diameters of target lesions, for small lymph nodes measuring <15 mm post therapy, a minimum absolute increase of 5 mm and the longest diameter should exceed 15mm, or appearance of new lesions. An MRD negative status will be defined as all results from whole blood and bone marrow that are negative for the presence of residual clonal cells (with assay sensitivity of 10^-6) per Adaptive Biotechnologies' reporting methods.
Time Frame: 2 years after date of BMT procedure for each patient
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Acalabrutinib
Number analyzed (Participants) | 15
percentage of participants
  PFS Rate Estimate of MRD-Negative Participants: number analyzed (Participants) | 12
  PFS Rate Estimate of MRD-Negative Participants | 88.9 [43.3 to 98.4]
  PFS Rate Estimate of MRD-Positive Participants: number analyzed (Participants) | 3
  PFS Rate Estimate of MRD-Positive Participants | 37.5 [1.1 to 80.8]

4. Secondary Outcome: Incidence of Grade 3 or Greater Treatment-Related Adverse Events
Description: Number of participants with grade 3 or higher CTCAE Version 5.0 Adverse Events that are considered related to study drug
Time Frame: Safety assessment will be done every cycle up to 2 years post-BMT
Population: All participants who have received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Acalabrutinib
Number analyzed (Participants) | 15
Participants | 6

ADVERSE EVENTS:
Time Frame: Serious and/or other adverse events were assessed from the date of first dose to 30 days after last dose of study treatment, up to 2 years post-BMT procedure. All-Cause Mortality was monitored from date of consent up to 5 years post-BMT procedure. This study closed early so full follow-up not collected for all patients so All-Cause Mortality was collected for a maximum of 3.7 years.
Description: All patients who received at least one dose of protocol treatment were followed for safety. Adverse events and serious adverse events were graded according to National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (NCI CTCAE) v5.0.
Groups:
- Acalabrutinib: Acalabrutinib will be self-administered orally for up to approximately 2 years post-BMT.
  Acalabrutinib: Acalabrutinib 129 mg BID will be self-administered orally starting from 100 day (+/- 7 days) Post-BMT on a 28-day schedule, until the patient has reached approximately 2 years post-BMT.
Arm/Group | Acalabrutinib
All-Cause Mortality (participants affected / at risk) | 0/15
Serious Adverse Events (participants affected / at risk) | 3/15
Other Adverse Events (participants affected / at risk) | 15/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Acalabrutinib (N=15)
Coronavirus infection (Infections and infestations) | 1
Clostridium difficile infection (Infections and infestations) | 1
Sepsis (Infections and infestations) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Acalabrutinib (N=15)
Anaemia (Blood and lymphatic system disorders) | 2
Neutropenia (Blood and lymphatic system disorders) | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 2
Lymphadenopathy (Blood and lymphatic system disorders) | 1
Palpitations (Cardiac disorders) | 1
Heart Rate Increased (Cardiac disorders) | 1
Ear Discomfort (Ear and labyrinth disorders) | 1
Ear Pruritus (Ear and labyrinth disorders) | 1
Hypoacusis (Ear and labyrinth disorders) | 1
Vertigo (Ear and labyrinth disorders) | 1
Hypothyroidism (Endocrine disorders) | 1
Androgen Deficiency (Endocrine disorders) | 1
Photophobia (Eye disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 8
Nausea (Gastrointestinal disorders) | 4
Abdominal Distension (Gastrointestinal disorders) | 2
Abdominal Pain (Gastrointestinal disorders) | 1
Abdominal Pain Upper (Gastrointestinal disorders) | 1
Anal Incontinence (Gastrointestinal disorders) | 1
Colitis (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 1
Oesophagitis (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Fatigue (General disorders) | 9
Pyrexia (General disorders) | 2
Chills (General disorders) | 1
Malaise (General disorders) | 1
Pain (General disorders) | 1
Oedema (General disorders) | 1
Covid-19 (Infections and infestations) | 4
Upper Respiratory Tract Infection (Infections and infestations) | 2
Eye Infection (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Sars-Cov-2 Test Positive (Infections and infestations) | 2
Bronchitis (Infections and infestations) | 1
Clostridium Difficile Infection (Infections and infestations) | 1
Coronavirus Infection (Infections and infestations) | 1
Exposure To Sars-Cov-2 (Infections and infestations) | 1
Gastroenteritis Viral (Infections and infestations) | 1
Influenza (Infections and infestations) | 1
Pharyngitis (Infections and infestations) | 1
Sepsis (Infections and infestations) | 1
Contusion (Injury, poisoning and procedural complications) | 1
Fall (Injury, poisoning and procedural complications) | 1
Spinal Compression Fracture (Injury, poisoning and procedural complications) | 1
Neutrophil Count Decreased (Investigations) | 3
Blood Creatinine Increased (Investigations) | 2
Weight Decreased (Investigations) | 2
Aspartate Aminotransferase Increased (Investigations) | 1
Blood Alkaline Phosphatase Increased (Investigations) | 1
Lymphocyte Count Decreased (Investigations) | 1
White Blood Cell Count Decreased (Investigations) | 1
Blood Uric Acid Increased (Investigations) | 1
Weight Increased (Investigations) | 1
Decreased Appetite (Metabolism and nutrition disorders) | 2
Dehydration (Metabolism and nutrition disorders) | 1
Hyperuricaemia (Metabolism and nutrition disorders) | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1
Vitamin D Deficiency (Metabolism and nutrition disorders) | 1
Vitamin B12 Deficiency (Metabolism and nutrition disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 4
Myalgia (Musculoskeletal and connective tissue disorders) | 4
Bone Pain (Musculoskeletal and connective tissue disorders) | 2
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 1
Neck Pain (Musculoskeletal and connective tissue disorders) | 1
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 1
Limb Injury (Musculoskeletal and connective tissue disorders) | 1
Headache (Nervous system disorders) | 6
Dizziness (Nervous system disorders) | 2
Peripheral Sensory Neuropathy (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 1
Aphasia (Nervous system disorders) | 1
Insomnia (Psychiatric disorders) | 2
Dysuria (Renal and urinary disorders) | 1
Acute Kidney Injury (Renal and urinary disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 2
Sinus Congestion (Respiratory, thoracic and mediastinal disorders) | 2
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 1
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea Exertional (Respiratory, thoracic and mediastinal disorders) | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Lower Respiratory Tract Congestion (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory Tract Congestion (Respiratory, thoracic and mediastinal disorders) | 1
Upper-Airway Cough Syndrome (Respiratory, thoracic and mediastinal disorders) | 1
Petechiae (Skin and subcutaneous tissue disorders) | 2
Rash (Skin and subcutaneous tissue disorders) | 2
Rash Maculo-Papular (Skin and subcutaneous tissue disorders) | 2
Dry Skin (Skin and subcutaneous tissue disorders) | 1
Nail Disorder (Skin and subcutaneous tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1
Basal Cell Carcinoma (Skin and subcutaneous tissue disorders) | 1
Dermatitis Acneiform (Skin and subcutaneous tissue disorders) | 1
Increased Tendency To Bruise (Skin and subcutaneous tissue disorders) | 1
Rash Pruritic (Skin and subcutaneous tissue disorders) | 1
Skin Lesion (Skin and subcutaneous tissue disorders) | 1
Squamous Cell Carcinoma (Skin and subcutaneous tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-09-29): https://cdn.clinicaltrials.gov/large-docs/38/NCT04402138/Prot_SAP_000.pdf